CLINICAL TRIAL: NCT01525290
Title: Efficacy and Safety of MRI-based Thrombolysis in Wake-up Stroke: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy and Safety of MRI-based Thrombolysis in Wake-up Stroke
Acronym: WAKE-UP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Götz Thomalla, MD, Coordinating Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WAKE-UP
Record Dates: First submitted 2012-01-30; First posted 2012-02-02 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Stroke
Keywords: wake-up stroke; thrombolysis; magnetic resonance imaging (MRI); diffusion weighted imaging (DWI); fluid attenuated inversion recovery (FLAIR)
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous tissue plasminogen activator (Experimental): Intervention drug: intravenous tissue plasminogen activator (tPA), alteplase
  Interventions: Drug: Alteplase
- Placebo (Placebo Comparator): Intervention drug: placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alteplase — Intravenous tissue plasminogen activator (Alteplase) 0.9 mg/kg body-weight up to a maximum of 90 mg, 10% as bolus, 90% over 1 hour as infusion
  Other Names: Actilyse; Activase; rt-PA
  Arms: intravenous tissue plasminogen activator
Drug: Placebo — lyophilised powder to be reconstituted as solution indistinguishable from the active drug
  Arms: Placebo

SUMMARY:
WAKE-UP is an investigator initiated European multicenter randomized controlled clinical trial of MRI based thrombolysis in acute stroke patients with unknown time of symptom onset, e.g. due to recognition of stroke symptoms on awakening. Objective of WAKE-UP is to prove efficacy and safety of MRI-based intravenous thrombolysis with Alteplase in patients waking up with stroke symptoms or patients with otherwise unknown symptom onset.

DETAILED DESCRIPTION:
WAKE-UP is a clinical trial of MRI based thrombolysis in acute stroke patients with unknown time of symptom onset, e.g. due to recognition of stroke symptoms on awakening. Intravenous thrombolysis with Alteplase is available as effective and safe treatment of acute stroke within 4.5 hours of symptom onset. However, in about 20% of acute stroke patients time of symptom onset is unknown. This large group of patients is currently excluded from treatment with Alteplase. The objective of the research proposed in the WAKE-UP project is to provide effective treatment options for this large group of acute stroke patients.

WAKE-UP is designed to prove efficacy and safety of MRI-based intravenous thrombolysis with Alteplase in patients waking up with stroke symptoms or patients with otherwise unknown symptom onset. Patients will be enrolled based on MRI findings indicative of acute ischemic stroke less than 4.5 hours of age.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria

* Clinical diagnosis of acute ischemic stroke with unknown symptom onset (e.g., stroke symptoms recognized on awakening)
* Last known well (without neurological symptoms) > 4.5 hours of treatment initiation
* Measurable disabling neurological deficit (defined as an impairment of one or more of the following: language, motor function, cognition, gaze, vision, neglect)
* Age 18-80 years
* Treatment can be started within 4.5 hours of symptom recognition (e.g., awakening)
* Written informed consent by patient or proxy

Imaging Inclusion Criteria:

* Acute stroke MRI including diffusion weighted imaging (DWI) and fluid attenuated inversion recovery (FLAIR) completed
* MRI showing a pattern of "DWI-FLAIR-mismatch", i.e. acute ischemic lesion visibly on DWI ("positive DWI") but no marked parenchymal hyperintensity visible on FLAIR ("negative FLAIR") indicative of an acute ischemic lesion ≤4.5 hours of age

Exclusion Criteria:

Clinical Exclusion Criteria

* Planned or anticipated treatment with endovascular reperfusion strategies (e.g. intra-arterial thrombolysis, mechanical recanalization techniques)
* Pre-stroke disability (inability to carry out all daily activities, requiring some help or supervision, i.e. slight disability corresponding to an MRS score > 1)
* Participation in any investigational study in the previous 30 days
* Severe stroke by clinical assessment (e.g. NIHSS > 25)
* Hypersensitivity to Alteplase or any of the excipients
* Pregnancy or lactating (formal testing needed in woman of childbearing potential; childbearing potential is assumed in women up to 55 years of age)
* Significant bleeding disorder at present or within past 6 months
* Known haemorrhagic diathesis
* Manifest or recent severe or dangerous bleeding
* Known history of or suspected intracranial haemorrhage
* Suspected subarachnoid haemorrhage (even if CT is negative) or condition after subarachnoid haemorrhage from aneurysm
* History of CNS damage (e.g. neoplasm, aneurysm, intracranial or spinal surgery)
* Recent (within 10 days) traumatic external heart massage, obstetrical delivery, recent puncture of a non-compressible blood-vessel
* Current use of anticoagulants (e.g. Phenprocoumon, Warfarin, new anticoagulants such as Dabigatran) or current use of heparin and elevated thromboplastin time (low-dose subcutaneous heparin is allowed)
* Platelet count < 100.000/mm3 (<100G/l)
* Blood glucose < 50 or > 400 mg/dl (< 2.8 or 22.2 mmol/l)
* Severe uncontrolled hypertension, i.e. systolic blood pressure > 185 mmHg or diastolic blood pressure >110 mmHg or requiring aggressive medication to maintain blood pressure within these limits (routine medical treatment is allowed to lower the blood pressure below these limits)
* Manifest or recent bacterial endocarditis, pericarditis
* Manifest or recent acute pancreatitis
* Documented ulcerative gastrointestinal disease during the last 3 months, oesophageal varices, arterial aneurysm, arterial/venous malformations
* Neoplasm with increased bleeding risk
* Manifest severe liver disease including hepatic failure, cirrhosis, portal hypertension and active hepatitis
* Major surgery or significant trauma in past 3 months
* Stroke within 30 days
* Life expectancy 6 months or less by judgement of the investigator
* Any condition associated with a significantly increased risk of severe bleeding not mentioned above
* Any contraindication to MRI (e.g. cardiac pacemaker)

Imaging Exclusion Criteria:

* Poor MRI quality precluding interpretation according to the study protocol
* Any sign of intracranial haemorrhage on baseline MRI
* FLAIR showing a marked parenchymal hyperintensity in a region corresponding to the acute DWI lesion indicative of an acute ischemic lesion with a high likelihood of being > 4.5 hours old
* Large DWI lesion volume > 1/3 of the MCA or > 50% of the anterior cerebral artery (ACA) or posterior cerebral artery (PCA) territory (visual inspection) or > 100 ml
* Any MRI findings indicative of a high risk of symptomatic intracranial haemorrhage related to potential IV-tPA treatment in the judgement of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Efficacy | 90 day after stroke
  Favourable outcome (Modified Rankin Scale 0-1)
Safety | 90 day after stroke
  * Mortality
  * Death or dependency (Modified Rankin Scale 4-6)

SECONDARY OUTCOMES:
Efficacy | 90 days after stroke
  * Global outcome score
  * Responder analysis (Modified Rankin Scale 0, 0-1 or 0-2 depending on severity of symptoms assessed by the National Institutes of Health Stroke Scale on admission)
  * Outcome across all disability ranges (categorical shift in Modified Rankin Scale score)
  * Infarct volume (measured 22-36 hours after treatment)
  * Functional health status and quality of life
  * Use of health care system resources
Safety | 90 days after stroke
  * Symptomatic intracranial haemorrhage (SICH) as defined in SITS-MOST
  * SICH as defined ECASS II
  * SICH as defined in NINDS
  * Parenchymal haemorrhage type 2 (PH-2)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gerloff, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Goetz Thomalla, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (7):
- Katholieke Universitet Leuven, Leuven, Belgium
- Aarhus Universitetshospital, Aahrhus Sygehus, Aarhus, Denmark
- Hospices Civils de Lyon, Bron, France
- Germany (2):
  - Charite - Universitätsmedizin Berlin, Berlin
  - University Medical Center Hamburg-Eppendorf, Hamburg
- Institut d'Investigacio Biomedica de Girona Doctor Josep Trueta, Girona, Spain
- University of Glasgow, Glasgow, United Kingdom

REFERENCES:
- [Result] Thomalla G, Simonsen CZ, Boutitie F, Andersen G, Berthezene Y, Cheng B, Cheripelli B, Cho TH, Fazekas F, Fiehler J, Ford I, Galinovic I, Gellissen S, Golsari A, Gregori J, Gunther M, Guibernau J, Hausler KG, Hennerici M, Kemmling A, Marstrand J, Modrau B, Neeb L, Perez de la Ossa N, Puig J, Ringleb P, Roy P, Scheel E, Schonewille W, Serena J, Sunaert S, Villringer K, Wouters A, Thijs V, Ebinger M, Endres M, Fiebach JB, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Gerloff C; WAKE-UP Investigators. MRI-Guided Thrombolysis for Stroke with Unknown Time of Onset. N Engl J Med. 2018 Aug 16;379(7):611-622. doi: 10.1056/NEJMoa1804355. Epub 2018 May 16. PMID 29766770
- [Derived] Nagele FL, Scheldeman L, Wouters A, Heinze M, Petersen M, Schlemm E, Schell M, Ebinger M, Endres M, Fiebach JB, Fiehler J, Galinovic I, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Puig J, Simonsen CZ, Thijs V, Thomalla G, Cheng B. Blood-Brain Barrier Leakage in the Penumbra Is Associated With Infarction on Follow-Up Imaging in Acute Ischemic Stroke. Stroke. 2025 Jul;56(7):1832-1842. doi: 10.1161/STROKEAHA.124.050171. Epub 2025 Apr 17. PMID 40242873
- [Derived] Galinovic I, Fiebach JB, Boutitie F, Cheng B, Cho TH, Ebinger M, Endres M, Enzinger C, Fiehler J, Ford I, Gregori J, Gunther M, Lemmens R, Muir KW, Nighoghossian N, Roy P, Simonsen CZ, Thijs VN, Wouters A, Gerloff C, Thomalla G, Pedraza S; for WAKE-UP Investigators. Effect of IV Thrombolysis With Alteplase in Patients With Vessel Occlusion in the WAKE-UP Trial. Neurology. 2025 Jan 28;104(2):e209871. doi: 10.1212/WNL.0000000000209871. Epub 2024 Dec 20. PMID 39705631
- [Derived] Frey BM, Shenas F, Boutitie F, Cheng B, Cho TH, Ebinger M, Endres M, Fiebach JB, Fiehler J, Galinovic I, Barow E, Konigsberg A, Schlemm E, Pedraza S, Lemmens R, Thijs V, Muir KW, Nighoghossian N, Simonsen CZ, Gerloff C, Thomalla G; WAKE-UP Investigators. Intravenous Thrombolysis in Patients With White Matter Hyperintensities in the WAKE-UP Trial. Stroke. 2023 Jul;54(7):1718-1725. doi: 10.1161/STROKEAHA.122.040247. Epub 2023 May 25. PMID 37226772
- [Derived] Jensen M, Sehner S, Cheng B, Schlemm E, Quandt F, Barow E, Wegscheider K, Boutitie F, Ebinger M, Endres M, Fiebach JB, Thijs V, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Simonsen CZ, Thomalla G, Gerloff C. Patient-Reported Quality of Life After Intravenous Alteplase for Stroke in the WAKE-UP Trial. Neurology. 2023 Jan 10;100(2):e154-e162. doi: 10.1212/WNL.0000000000201375. Epub 2022 Oct 27. PMID 36302662
- [Derived] Barow E, Quandt F, Cheng B, Gelderblom M, Jensen M, Konigsberg A, Boutitie F, Nighoghossian N, Ebinger M, Endres M, Fiebach JB, Thijs V, Lemmens R, Muir KW, Pedraza S, Simonsen CZ, Gerloff C, Thomalla G. Association of White Blood Cell Count With Clinical Outcome Independent of Treatment With Alteplase in Acute Ischemic Stroke. Front Neurol. 2022 Jun 13;13:877367. doi: 10.3389/fneur.2022.877367. eCollection 2022. PMID 35769368
- [Derived] Schlemm L, Braemswig TB, Boutitie F, Vynckier J, Jensen M, Galinovic I, Simonsen CZ, Cheng B, Cho TH, Fiehler J, Puig J, Thijs V, Fiebach J, Muir K, Nighoghossian N, Ebinger M, Pedraza S, Thomalla G, Gerloff C, Endres M, Lemmens R, Nolte CH; WAKE-UP Investigators. Cerebral Microbleeds and Treatment Effect of Intravenous Thrombolysis in Acute Stroke: An Analysis of the WAKE-UP Randomized Clinical Trial. Neurology. 2022 Jan 18;98(3):e302-e314. doi: 10.1212/WNL.0000000000013055. Epub 2021 Nov 15. PMID 34782419
- [Derived] Lettow I, Jensen M, Schlemm E, Boutitie F, Quandt F, Cheng B, Ebinger M, Endres M, Fiebach JB, Thijs V, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Simonsen CZ, Gerloff C, Thomalla G; WAKE-UP Investigators. Serious Adverse Events and Their Impact on Functional Outcome in Acute Ischemic Stroke in the WAKE-UP Trial. Stroke. 2021 Dec;52(12):3768-3776. doi: 10.1161/STROKEAHA.120.033425. Epub 2021 Aug 26. PMID 34433305
- [Derived] Barow E, Boutitie F, Cheng B, Cho TH, Ebinger M, Endres M, Fiebach JB, Fiehler J, Nickel A, Puig J, Roy P, Lemmens R, Thijs V, Muir KW, Nighoghossian N, Pedraza S, Simonsen CZ, Gerloff C, Thomalla G. 24-hour blood pressure variability and treatment effect of intravenous alteplase in acute ischaemic stroke. Eur Stroke J. 2021 Jun;6(2):168-175. doi: 10.1177/23969873211014758. Epub 2021 Jun 18. PMID 34414292
- [Derived] Scheldeman L, Wouters A, Dupont P, Christensen S, Boutitie F, Cheng B, Ebinger M, Endres M, Fiebach JB, Gerloff C, Muir KW, Nighoghossian N, Pedraza S, Simonsen CZ, Ringelstein EB, Chamorro A, Grond M, Laage R, Schneider A, Thomalla G, Thijs V, Lemmens R. Reversible Edema in the Penumbra Correlates With Severity of Hypoperfusion. Stroke. 2021 Jul;52(7):2338-2346. doi: 10.1161/STROKEAHA.120.033071. Epub 2021 May 13. PMID 33980046
- [Derived] Konigsberg A, Sehner S, Arlt S, Cheng B, Simonsen CZ, Boutitie F, Serena J, Thijs V, Ebinger M, Endres M, Fiebach JB, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Gerloff C, Thomalla G; WAKE-UP investigators. Effect of intravenous alteplase on post-stroke depression in the WAKE UP trial. Eur J Neurol. 2021 Jun;28(6):2017-2025. doi: 10.1111/ene.14797. Epub 2021 Mar 22. PMID 33657675
- [Derived] Grosch AS, Kufner A, Boutitie F, Cheng B, Ebinger M, Endres M, Fiebach JB, Fiehler J, Konigsberg A, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Siemonsen CZ, Thijs V, Wouters A, Gerloff C, Thomalla G, Galinovic I. Extent of FLAIR Hyperintense Vessels May Modify Treatment Effect of Thrombolysis: A Post hoc Analysis of the WAKE-UP Trial. Front Neurol. 2021 Feb 4;11:623881. doi: 10.3389/fneur.2020.623881. eCollection 2020. PMID 33613422
- [Derived] Barow E, Pinnschmidt H, Boutitie F, Konigsberg A, Ebinger M, Endres M, Fiebach JB, Fiehler J, Thijs V, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Simonsen CZ, Gerloff C, Thomalla G, Cheng B; WAKE-UP investigators. Symptoms and probabilistic anatomical mapping of lacunar infarcts. Neurol Res Pract. 2020 Aug 3;2:21. doi: 10.1186/s42466-020-00068-y. eCollection 2020. PMID 33324925
- [Derived] Schlemm L, Kufner A, Boutitie F, Nave AH, Gerloff C, Thomalla G, Simonsen CZ, Ford I, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Ebinger M, Endres M. Current Smoking Does Not Modify the Treatment Effect of Intravenous Thrombolysis in Acute Ischemic Stroke Patients-A Post-hoc Analysis of the WAKE-UP Trial. Front Neurol. 2019 Nov 22;10:1239. doi: 10.3389/fneur.2019.01239. eCollection 2019. PMID 31824412
- [Derived] Barow E, Boutitie F, Cheng B, Cho TH, Ebinger M, Endres M, Fiebach JB, Fiehler J, Ford I, Galinovic I, Nickel A, Puig J, Roy P, Wouters A, Thijs V, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Simonsen CZ, Gerloff C, Thomalla G; WAKE-UP investigators. Clinical Characteristics and Outcome of Patients with Lacunar Infarcts and Concurrent Embolic Ischemic Lesions. Clin Neuroradiol. 2020 Sep;30(3):511-516. doi: 10.1007/s00062-019-00800-5. Epub 2019 Jun 3. PMID 31161343
- [Derived] Thomalla G, Boutitie F, Fiebach JB, Simonsen CZ, Nighoghossian N, Pedraza S, Lemmens R, Roy P, Muir KW, Heesen C, Ebinger M, Ford I, Cheng B, Cho TH, Puig J, Thijs V, Endres M, Fiehler J, Gerloff C. Effect of informed consent on patient characteristics in a stroke thrombolysis trial. Neurology. 2017 Sep 26;89(13):1400-1407. doi: 10.1212/WNL.0000000000004414. Epub 2017 Aug 25. PMID 28842449
- [Derived] Thomalla G, Boutitie F, Fiebach JB, Simonsen CZ, Pedraza S, Lemmens R, Nighoghossian N, Roy P, Muir KW, Ebinger M, Ford I, Cheng B, Galinovic I, Cho TH, Puig J, Thijs V, Endres M, Fiehler J, Gerloff C. Clinical characteristics of unknown symptom onset stroke patients with and without diffusion-weighted imaging and fluid-attenuated inversion recovery mismatch. Int J Stroke. 2018 Jan;13(1):66-73. doi: 10.1177/1747493017706245. Epub 2017 Apr 20. PMID 28425349
- [Derived] Thomalla G, Boutitie F, Fiebach JB, Simonsen CZ, Nighoghossian N, Pedraza S, Lemmens R, Roy P, Muir KW, Ebinger M, Ford I, Cheng B, Galinovic I, Cho TH, Puig J, Thijs V, Endres M, Fiehler J, Gerloff C; WAKE-UP Investigators. Stroke With Unknown Time of Symptom Onset: Baseline Clinical and Magnetic Resonance Imaging Data of the First Thousand Patients in WAKE-UP (Efficacy and Safety of MRI-Based Thrombolysis in Wake-Up Stroke: A Randomized, Doubleblind, Placebo-Controlled Trial). Stroke. 2017 Mar;48(3):770-773. doi: 10.1161/STROKEAHA.116.015233. Epub 2017 Feb 7. PMID 28174327